CLINICAL TRIAL: NCT00203970
Title: Diffusion of Use of Low Molecular Weight Heparin for Thrombosis on the Medicine Services
Status: Active, not recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10895A
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Thrombosis
Keywords: Thrombosis; Low Molecular Weight Heparin
MeSH Terms: conditions — Thrombosis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Observation — Using a data abstraction form, we wish to gather the following information: 1) Patient demographics 2) identity of the attending, residents, and interns caring for the patient 3)whether the patient had any absolute or relative contraindications for receiving LMWH 4) how the patient was treated for his/her condition

SUMMARY:
The purpose of this research is to gain insight into the way in which physicians adopt new practice techniques. In particular, we are interested in how medical innovations diffuse throughout social networks. We wish to examine the diffusion of Low Molecular Weight Heparin (LMWH) use for Deep Vein Thrombosis (DVT) throughout the social network of general internal medicine interns, residents, and attendings at the University of Chicago Hospital. In numerous clinical trials, LMWH has been demonstrated to be as effective as unfractionated heparin as a bridge to long-term anticoagulation therapy with Coumadin, with the added benefit of early discharge from the hospital with easy dosing, no need for monitoring, and home therapy. A DVT critical pathway was established at the U of C in 1998, and LMWH was used off-label for that purpose beginning in 1997. However, it is unclear how quickly the use of LMWH was adopted by the physicians on the general medicine services, or whether there exists a pattern for this adoption.

DETAILED DESCRIPTION:
The design of our study is retrospective in nature. We are interested primarily in the use of LMWH in patients admitted to the general medicine services between January 1, 1997 and February 1, 2001 with a primary and secondary diagnosis related to Venous Thromboembolism, including specific ICD-9 codes.

Using a data abstraction form, we gather the following information: 1) patient demographics, 2) identity of the attending, resident, and interns caring for the patient, 3) whether the patient had any absolute or relative contraindications for receiving LMWH, as delineated by the DVT critical pathway, including insurance status and 4)how the patient was treated for his/her condition. To examine whether the identity of the primary care physician affects whether LMWH is given, we also collect the name of the primary care physician if it is listed on the chart.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to General Medicine Services with a primary or secondary diagnosis related to venous thromboembolism

Exclusion Criteria:

* Non-General Medicine Services patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted into the general medicine services with a primary or secondary diagnosis related to Venous Thromboembolism.
Sampling Method: Probability Sample
Enrollment: 645 (Actual)
Dates: Start 2001-02; Primary Completion 2001-03 (Actual); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
retrospective chart review to determine how patients with deep venous thromboses or pulmonary emboli were treated when hospitalized on the medicine services | June 1997 to December 2000
  Using the data abstraction form, we gathered the following information: 1) patient demographics, 2) the identity of the attending, resident, and intern caring for the patient, 3) whether the patient had any absolute or relative contraindications for receiving LMWH, as delineated by the DVT critical pathway, including insurance status and 4) how the patient was treated for his/her condition.

CONTACTS AND LOCATIONS:
Overall Officials: David Meltzer, M.D., Ph.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States